CLINICAL TRIAL: NCT03612154
Title: A Phase II Study of Lorlatnib in ROS1 Rearranged Advanced NSCLC
Brief Title: Study of Lorlatinib in ROS1 Rearranged NSCLC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Cancer Center, Korea (Other Government)
Responsible Party: Principal Investigator, Ji-youn Han, MD. PhD., National Cancer Center, Korea
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCC-2018-0232
Record Dates: First submitted 2018-06-14; First posted 2018-08-02 (Actual); Last update posted 2022-04-06 (Actual); Status verified 2022-04

CONDITIONS: Nonsmall Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — lorlatinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Lorlatinib (Experimental): Subjects will be treated with lorlatinib 100mg PO daily. A cycle will be defined as 28-days for the convenience of analysis.
  Interventions: Drug: Lorlatinib

INTERVENTIONS:
Drug: Lorlatinib — Subjects will be treated with lorlatinib 100mg PO daily. A cycle will be defined as 28-days for the convenience of analysis.

SUMMARY:
This is a phase II, multi-center, single arm study of lorlarinib as a single agent in patients with ROS1-rearranged advanced NSCLC.

DETAILED DESCRIPTION:
ROS1 rearrangement characterizes a small subset (1-2%) of non-small cell lung cancer (NSCLC) and is associated with light or never smoking patients and adenocarcinoma histology. Recently, ROS1 inhibitors such as crizotinib and ceritinib demonstrated significant efficacy in ROS1 rearranged NSCLC. Thus, identification of ROS1 rearrangement in NSCLC is mandatory to permit ROS1 targeted therapy. However, current guidelines either do not refer to ROS1 testing or mention it briefly without making any strong recommendation. The detection of ROS1rearrangement is based on in situ (immunohistochemistry [IHC], fluorescence in situ hybridization [FISH]) and extractive non-in situ assays. While FISH still represents the gold standard in clinical trials, this technique may fail to recognize rearrangements of ROS1 with some gene fusion partner. On the other hand, IHC is the most cost-effective screening technique, but it seems to be characterized by low specificity. Extractive molecular assays are expensive and laborious methods, but they specifically recognize almost all ROS1 fusions using a limited amount of mRNA even from formalin-fixed, paraffin-embedded tumor tissues. Recently, Korean Heath Insurance Review and Assessment Service (HIRA) approved next generation sequencing (NGS)-based target sequencing for NSCLC patients, which may facilitate the detection of ROS1 rearrangement in Korean patients with advanced NSCLC.

Lorlatinib is a new, potent, brain-penetrant, ATP-competitive small molecule inhibiter of ALK/ROS1. However, the objective response rate (ORR) was 17/47 (36.2%; 95% CI 22.7, 51.5) in ROS1 arm of B7461001 study, but this result may not represent the ORR of lorlatinib as a 1st line treatment since 53% had central nervous system involvement at baseline and 72% of patients had received prior crizotinib. Therefore, given the activity of lorlatinib in ROS1 rearranged lung cancer, The investigator will investigate the efficacy of lorlatinib in ROS1 inhibitor-naïve patients with ROS1- rearranged NSCLC. The investigator will also investigate the efficacy according to fusion partners and resistance mechanisms. Finally, The investigator will compare the concordance among diagnostic tests including FISH, IHC and NGS-based target sequencing and provide the clinical guidance for diagnosis of ROS1 rearrangement in NSCLC.

ELIGIBILITY:
4.1. Inclusion criteria

1. Metastatic or recurrent NSCLC with ROS1 rearrangement identified by NGS-based target sequencing
2. Treatment naïve or one prior systemic treatment with platinum doublet chemotherapy
3. At least one measurable disease lesion according to RECIST 1.1
4. ECOG performance status 0-2
5. Age ≥ 18 years
6. Adequate hematologic, hepatic, and renal function
7. Written informed consent

4.2. Exclusion criteria

1. Life expectancy of less than 12 weeks
2. Prior treatment with a ROS1 inhibitor
3. Symptomatic uncontrolled brain metastasis
4. Other malignancy within 5 years, except for adequately treated carcinoma in situ of the cervix, basal or squamous cell skin cancer, localized prostate cancer treated surgically with curative intent, and ductal carcinoma in situ treated surgically with curative intent
5. Uncontrolled intercurrent illness
6. Pregnancy or unwillingness to use effective birth control
7. Known hypersensitivity to lorlatinib and/or its excipients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2019-05-02 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
ORR | from Cycle1 Day 1 until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months").
  To assess the clinical efficacy of lorlatinib as measured by ORR using RECIST criteria v 1.1

CONTACTS AND LOCATIONS:
Overall Officials: Ji-Youn Han, MD.Ph.D., Principal Investigator — National Cancer Center
Locations (1):
- National Cancer Center, Goyang-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ahn BC, Kim YJ, Lee Y, Suh KJ, Kim SH, Kim DW, Kim TM, Lee KH, Han JY. Lorlatinib in Tyrosine Kinase Inhibitor-Naive Advanced ROS1-Positive Non-Small Cell Lung Cancer: A Phase 2 Nonrandomized Clinical Trial. JAMA Oncol. 2026 Jan 1;12(1):84-89. doi: 10.1001/jamaoncol.2025.5097. PMID 41296331